CLINICAL TRIAL: NCT06334263
Title: Decision to Treat Acute Traumatic Splenic Artery Injury in the Context of Trauma
Brief Title: Splenic Embolisation Decisions
Acronym: SPEED
Status: Recruiting | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 332302
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Trauma; Spleen Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conservative management: No intervention for splenic injury other than supportive care
- Splenic embolisation: Interventional radiology guided splenic artery embolisation
- Splenectomy: Surgical splenectomy

SUMMARY:
The spleen is often injured when the body sustains trauma. This leads to bleeding. The bleeding can be stopped by a big operation cutting open the belly or a small hole in your groin where a blood vessel can be accessed and through which the bleeding can be stopped. We do not know what types of injuries it is best to use this procedure. We do not know why we do not use the smaller technique in some instances. We also do not know exactly which of a number of ways to stop the bleeding could be better. We have a big data set in the trauma and audit research network (TARN) which we would like to use to help answer these questions and design further studies to better answer the questions. Adding a few other pieces of data, we are able to answer key questions into how the spleen will best be treated in trauma.

DETAILED DESCRIPTION:
Splenic embolisation (SE) is a minimally invasive procedure whereby the splenic artery is blocked to stop bleeding from the spleen. This is typically undertaken in the context of acute traumatic splenic injury, diagnosed using Computed Tomography (CT) Scan by a diagnostic radiologist. The vessel can be accessed using wires and catheters under imaging guidance with access typically though the common femoral artery. This has been shown to be a viable management option in patients who are traumatically injured, in the absence of concurrent immediately life-threatening other injuries requiring damage control surgery (DCS).

Splenic injury is classified according to the American Association of Trauma Surgery (AAST) grade (grades 1 to 5), with increased severity traumatic injury according to the higher numerical value. SE is typically performed in higher grade (3/4) splenic injuries, although the gold standard of management of Grade 5 is considered surgical resection. There is no current definitive consensus as to appropriateness of the management of these grades although there is a trend towards embolisation since the inception of trauma networks in England in 2012. The 22 Trauma centres now function as a hub for trauma within their specified area and had the aim of developing trauma services and improving clinical care. The 22 Adult Trauma centres within England are listed in appendix A. There are few guidelines regarding the availability and specifications of interventional radiology (IR) provision at Major Trauma Centres (MTCs) and there is no available data on the impact of IR on-call structure and quality or location of IR facilities on the splenic conservation rate and time to treatment. SE technique and rate are variable and depend on multiple factors. These factors include the time to CT report, the availability of On Call IR services, the method of contact of the IR, availability of a hybrid theatre and the associated injuries. A recent survey of British Society of Interventional Radiology (BSIR) members, undertaken as part of the BSIR audit and registry committee, demonstrated wide variability in the management and treatment of splenic injuries with respect to SE (unpublished data). This was due to a number of factors regarding service design and decisions around appropriateness and method of embolisation. Splenic embolisation can be performed in two main ways, either with a proximal occlusion of the splenic artery outside of its hilum, or within the actual splenic tissue having selected the arterial branch that is demonstrated as bleeding. The embolisation (stopping of the bleeding) can be performed using a variety of methods, including coils, plugs, gelfoam or glue to stop the blood getting to the damaged vessel. The technique and method of embolisation also have a poor evidence base. No multicentre UK based dataset has been published. This highlights the lack of consensus, guidelines, and research in this area. Work on the available retrospective dataset which are available through Trauma and Audit Research Network (TARN) should be undertaken to analyse the current situation to enable design of multi-centre prospective research. This work will benefit patients by establishing an improved evidence base regarding the optimum service design and treatment pathway. We aim to benefit the NHS by clearly identifying factors that improve the successful embolisation rate, a less invasive procedure than damage control surgery (DCS) whereby a surgeon would remove the spleen through a large incision in the abdomen. We aim to clarify the role of and support the development of IR within the trauma setting by establishing a more evidence-based practice to support interventional radiologists in their decision-making around splenic embolisation in the context of Acute Traumatic Splenic injury (ATSI). The determination of the impact IR service design on outcomes will enable improved management decisions on overall patient care.

ELIGIBILITY:
INCLUSION Criteria:

All patients who had traumatic splenic injury between 01/01/2016 and 31/12/2020 with data available from TARN CT available for review.

EXCLUSION CRITERIA:

CT not available to radiologically grade the Splenic injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients identified as having an acute traumatic splenic injury grade AAST 2-5 on the TARN database between the given dates will be included. Hospitals who decline participation in the data collection will have their patients excluded from the analysis excluded by site as identified in TARN database
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Splenic embolisation rate as percentage of; acute splenic trauma per Major Trauma Centre (MTC) | 5 years
  Splenic embolisation rate as percentage of; acute splenic trauma, per injury grade and per Major Trauma Centre (MTC). Failure of conservative management rate and splenectomy rate.
Number of On call IR consultants affecting embolisation rate | 5 years
  Does the number of on call IR consultants affect the embolisaiton rate
What is the splenic salvage rate for proximal versus distal embolisation | 5 years
  What is the splenic salvage rate for proximal versus distal embolisation
Readmission rate of splenic embolisation versus splenectomy | 5 years
  Readmission rate of splenic embolisation versus splenectomy
Embolisation failure | 5 years
  Embolisation failure rate

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Plymouth NHS Trust, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chakraverty S, Flood K, Kessel D, McPherson S, Nicholson T, Ray CE Jr, Robertson I, van Delden OM. CIRSE guidelines: quality improvement guidelines for endovascular treatment of traumatic hemorrhage. Cardiovasc Intervent Radiol. 2012 Jun;35(3):472-82. doi: 10.1007/s00270-012-0339-7. Epub 2012 Jan 20. No abstract available. PMID 22271075
- [Background] Kozar RA, Crandall M, Shanmuganathan K, Zarzaur BL, Coburn M, Cribari C, Kaups K, Schuster K, Tominaga GT; AAST Patient Assessment Committee. Organ injury scaling 2018 update: Spleen, liver, and kidney. J Trauma Acute Care Surg. 2018 Dec;85(6):1119-1122. doi: 10.1097/TA.0000000000002058. No abstract available. PMID 30462622
- [Background] Yiannoullou P, Hall C, Newton K, Pearce L, Bouamra O, Jenks T, Scrimshire AB, Hughes J, Lecky F, Macdonald A. A review of the management of blunt splenic trauma in England and Wales: have regional trauma networks influenced management strategies and outcomes? Ann R Coll Surg Engl. 2017 Jan;99(1):63-69. doi: 10.1308/rcsann.2016.0325. Epub 2016 Oct 28. PMID 27791418
- [Background] 4. RCR 2015 - Standards for practice and guidance for trauma radiology in the severely injured patient. Available at: https://www.rcr.ac.uk/system/files/publication/field_publication_files/bfcr155_traumaradiol.pdf
- [Background] Schnuriger B, Inaba K, Konstantinidis A, Lustenberger T, Chan LS, Demetriades D. Outcomes of proximal versus distal splenic artery embolization after trauma: a systematic review and meta-analysis. J Trauma. 2011 Jan;70(1):252-60. doi: 10.1097/TA.0b013e3181f2a92e. PMID 21217497
- [Background] Foley PT, Kavnoudias H, Cameron PU, Czarnecki C, Paul E, Lyon SM. Proximal Versus Distal Splenic Artery Embolisation for Blunt Splenic Trauma: What is the Impact on Splenic Immune Function? Cardiovasc Intervent Radiol. 2015 Oct;38(5):1143-51. doi: 10.1007/s00270-015-1162-8. Epub 2015 Jul 3. PMID 26139039